CLINICAL TRIAL: NCT07239544
Title: Generation of Tumor-reactive T Cells Based on Tumor Whole Cell Antigen Nanovaccines
Brief Title: Generation of Reactive T Cells Based on Tumor Whole Cell Antigen Nanovaccines
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025666
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — observational study:Evaluate the broad-spectrum coverage of xenogeneic hybrid lung cancer antigens (including patient tissues and cell lines), and develop a universal whole-cell antigen nanodelivery system to replace autologous tumor-derived preparation

SUMMARY:
Tumor-reactive T cells are generated based on the tumor full antigen nanovaccine and the tumor-reactive T cells are reinjected for autologous therapy to provide the optimal treatment plan for clinical patients.

DETAILED DESCRIPTION:
To evaluate the anti-tumor effect of tumor-reactive T cells in human-derived 3D lung cancer organoids, and analyze the in vivo migration location, tumor infiltration characteristics and survival kinetics of reinjected tumor-reactive T cells to clarify their role in biotherapy and transformation potential.

ELIGIBILITY:
Inclusion Criteria:

- a.Freshly frozen tumor tissue samples of at least 0.5cm*0.5cm in length and diameter were obtained from patients with histologically confirmed primary non-small cell lung cancer (NSCLC) who underwent surgical resection.

b. HLA typing must match the preselected subtypes: prioritize common subtypes such as HLA-A*0201 and HLA-A*2402 to ensure standardized subsequent T-cell response evaluation.

Exclusion Criteria:

- a.History of active autoimmune diseases: such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc., to avoid vaccine-induced immune storm.

b. Previous immunotherapy: including PD-1/L1 inhibitors, CTLA-4 inhibitors, cancer vaccines, or other cellular therapies within 6 months, with treatment interference excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient private information is kept confidential and shall not be disclosed publicly. The patient information is for research purposes only and shall not be used for any commercial purpose.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Tumor reactive cells | 6 month
  To evaluate the antitumor effects of tumor-reactive T cells in human 3D lung cancer organoids, and to elucidate the in vivo migration and localization, tumor infiltration characteristics, and survival dynamics of reinfused tumor-reactive T cells, thereby clarifying their role and translational potential in biological therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No